CLINICAL TRIAL: NCT00408226
Title: Phase 1/2 Study of Oral MKC-1 Administered Twice Daily for 14 Consecutive Days Every 3 Weeks in Combination With Pemetrexed
Brief Title: Safety Study of MKC-1 Combined With Pemetrexed to Treat Advanced Cancer and Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Chief Medical Officer, EntreMed, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKC-102
Record Dates: First submitted 2006-12-05; First posted 2006-12-06 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Advanced Cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MKC-1; Drug: pemetrexed

INTERVENTIONS:
Drug: MKC-1 — capsules, twice daily for 14 days in 21 day cycle
Drug: pemetrexed — standard dosing of 500 mg/m2 infused every 21 days

SUMMARY:
To determine the toxicities, maximum tolerated dose (MTD) and recommended phase 2 dose of MKC-1 when administered orally, twice daily for 14 days followed by 7 days without dosing, in combination with pemetrexed (delivered at its recommended single agent dose) to patients with advanced solid tumor malignancies. Also, to determine the antitumor activity, based on the objective response rate and median Progression Free Survival ("PFS"), of oral MKC-1, administered on this schedule in combination with pemetrexed to patients with non small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must satisfy this criteria based on the portion of the study for which they are being considered for enrollment:

   Dose Escalating Phase: Patients with advanced solid tumor malignancies for whom single-agent pemetrexed therapy would not be contraindicated. Measurable disease not required.

   Phase 2 portion: Current diagnosis of Stage IIIb (due to malignant pleural effusion or supraclavicular lymph node involvement only) or Stage IV histologically and/or cytologically proven non-small cell lung cancer according to staging system of the American Joint Committee on Cancer.

   (i) Patient has received maximally feasible surgical resection and/or radiotherapy for initial disease.

   (ii) Either disease progression following treatment with one prior chemotherapy regimen used for the treatment of metastatic disease or disease progression following adjuvant/neoadjuvant therapy within one year of last dose of chemotherapy or (for those patients with disease progression following adjuvant/neoadjuvant therapy >1 year of last dose of chemotherapy) disease progression following one additional chemotherapy regimen for metastatic disease.

   (iii) Radiographic or physical examination evidence of at least one site of unidimensionally-measurable disease, using the RECIST criteria with disease assessed within 28 days prior to treatment initiation.
2. Age ≥ 18 years.
3. ECOG performance status of 0 or 1.
4. All acute toxicity of any prior chemotherapy, surgery or radiotherapy must have resolved to NCI CTCAE Grade ≤ 1, except for alopecia.
5. The following laboratory results, within 10 days of MKC-1 administration:

   Hemoglobin ≥ 9 g/dL Absolute neutrophil count ≥ 1.5 x 109/L Platelet count ≥ 75 x 109/L Serum creatinine ≤ 1.5 x ULN (upper limit of normal) Creatinine clearance ≥ 45 mL/min AST ≤ 2.5 x ULN Serum albumin ≥ LLN (lower limit of normal) or 3.5 g/dL Total bilirubin ≤ ULN
6. Signed informed consent.

Exclusion Criteria:

1. Pre-existing hepatomegaly with disease measured as ≥ 2 cm below the costal margin, secondary to malignancy.
2. Uncontrolled pleural effusions (defined as more than 2 pleuracenteses within 4 weeks of the first dose of study drug)
3. Administration of cancer-specific therapy within the following periods prior to study drug initiation:

   * less than 4 weeks prior: major surgery (this does not include placement of venous access device or biopsy) or any investigational therapy;
   * less than 3 weeks prior: radiation therapy or chemotherapy (except for oral EGF-R receptor tyrosine kinase inhibitor(s);
   * less than 2 weeks prior: oral EGF-R receptor tyrosine kinase inhibitor(s).
4. Pregnant or breast-feeding women. Female patients must be postmenopausal, surgically sterile or they must agree to use a physical method of contraception. Female patient with childbearing potential must have a negative pregnancy test within the 10 days before the first MKC-1 administration. Male patients must be surgically sterile or agree to use an acceptable method of contraception.
5. Known CNS or leptomeningeal metastases unless treated, clinically stable and not requiring steroids.
6. Clinical evidence of bowel obstruction, active uncontrolled malabsorption syndromes or a history of total gastrectomy.
7. Uncontrolled hypercalcemia (serum calcium-corrected > 12 mg/dL)
8. Serious cardiac condition (Class III/IV congestive heart failure according to New York Heart Association classification); documented acute myocardial infarction within the previous 6 months.
9. Any medical conditions that, in the investigator's opinion, would impose excessive risk to the patient. Examples of such conditions include congestive heart failure of Class III or IV of the NYHA classification, infection requiring parenteral or oral anti-infective treatment, any altered mental status or any psychiatric condition that would interfere with the understanding of the informed consent.
10. Patients with active secondary malignancies.
11. Treatment with antiretroviral therapy metabolized through CYP3A4 (including indinavir, nelfinavir, ritonavir and saquinavir).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-10; Primary Completion 2009-06 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of treatment emergent AEs | throughout study participation

CONTACTS AND LOCATIONS:
Overall Officials: Nasser H. Hanna, M.D., Principal Investigator — Indiana University School of Medicine
Locations (4):
- United States (4):
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Swedish Cancer Institute, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin